CLINICAL TRIAL: NCT03322449
Title: APOA2 Gene, Diet, Inflammation and Gut Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Jose Ordovas, Senior Scientist, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-08911
Record Dates: First submitted 2017-09-08; First posted 2017-10-26 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Inflammation
Keywords: APOA2; Inflammation; gene; diet
MeSH Terms: conditions — Inflammation | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: randomized crossover dietary intervention
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal Diet (Experimental): during this Arm, the participants will receive a diet enriched in animal products
  Interventions: Other: Animal Diet
- Plant Diet (Experimental): during this Arm, the participants will receive a diet enriched in plant products
  Interventions: Other: Plant Diet

INTERVENTIONS:
Other: Animal Diet — during one week participants will receive food products enriched in animal products and with high content of fat and protein
  Arms: Animal Diet
Other: Plant Diet — during one week participants will receive plant products enriched in fiber and complex carbohydrates
  Arms: Plant Diet

SUMMARY:
Nutrients and chemicals in food are able to regulate expression of genetic elements. Gene-nutrient interaction in response to unhealthy diets can increase an individual's risk, shifting the individual from health toward the development of chronic disease. The apolipoprotein A2 (APOA2) gene may either put individuals at risk for or protect from obesity in the presence of certain fats in food. The main purpose of this four-week study is to examine diet induced gene-nutrient interaction, with a focus on gut health, gut microbiota and inflammation in individuals who have either the CC or the TT form within a specific variant of the APOA2 Gene. The (2) one-week study diets, one plant based and the other animal based are separated by a (1) week return to your regular habitual without probiotic or prebiotic food products.

DETAILED DESCRIPTION:
The primary objectives of this application are 1. To use a diet intervention setting to rigorously evaluate the mechanisms responsible for the previously observed effects, focusing on gut microbiota and markers of gut health and inflammation and 2. To prove that targeted dietary intervention based on genes can provide additional, tailored benefit to genetically vulnerable individuals. The overall hypothesis proposes that significant cross-talk between the human host genome, the microbiome, and the diet, defines the observed inter-individual variation in metabolic and physiological responses. Accordingly, the investigators propose the following specific aims and hypotheses.

AIM 1: To catalog the response of the plasma metabolome to diets differing in saturated fat and prebiotics content (animal-based diet versus plant-based diet) in individuals from the USA carrying CC (n=20) and TT (n=20) genotypes at the common APOA2 -265T>C SNP using a crossover, randomized dietary intervention study.

Our primary hypothesis states: A significant and biologically relevant proportion of the individual variation in changes in the plasma metabolome in response to dietary saturated fat and prebiotic intake will be due to APOA2-265T>C genotypes. Specifically, subjects homozygous (CC) for the less common C allele will respond to decreases in total dietary saturated fat and increases in prebiotics (i.e., plant-based diet) with significantly greater improvement of metabolites related to gut health, inflammation and other cardiometabolic traits than subjects homozygous (TT) for the common T allele.

AIM 2: To characterize differential impacts of low SFA/high prebiotic (plant-based) diet vs. high SFA/low prebiotic (animal-based) diets on gut microbiota patterns between CC and TT persons at APOA2-265T>C.

Our primary hypothesis states: CC subjects have a preference for high-fat and -protein foods and therefore high levels of Bacteroidetes, Actinobacteria and similar species in the gut are expected. Moreover, reducing intake of saturated fat and increasing prebiotics will be more effective in inducing a healthier gut microflora profile in CC subjects than in those with the TT genotype, with opposite effects observed when the diet is switched to one high in saturated fat.

AIM 3: To integrate the metabolomic and gut microflora taxonomic information generated in AIM1 and AIM2 in order to elucidate the physiological mechanism(s) by which diet impinges on metabolic pathways through APOA2 genotypes.

Our primary hypothesis states: A diet low in saturated fat and high in prebiotics induces beneficial changes in gut microbiota, metabolic processes and inflammation, which are significantly more pronounced in CC than in TT subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18 years or older
* Women who are not pregnant
* A BMI ranging between 27 and 34

Exclusion Criteria:

* Unexplained elevation in serum transaminases (i.e. >1.5 times the upper limit of normal) or with evidence of active liver disease, including primary biliary cirrhosis or pre-existing gallbladder disease
* Severe renal dysfunction (serum creatinine >2.0mg/dL)
* Excessive alcohol consumption (>2 drinks/day)
* Preexisting cardiovascular disease (CVD)
* Stable exertional angina pectoris requiring sublingual nitroglycerin within the prior 3 months
* Uncontrolled tyoe 2 diabetes (T2D) (fasting glucose >126 mg/dl) or other significant endocrine disease.
* Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg).
* History of pancreatitis within 1 yr. prior to screening.
* Subjects on lipid lowering or diabetes medications.
* Smoking
* Pregnancy
* Body mass index (BMI) below 27 or greater than 34 kg/m2
* Participants will also be excluded for drug abuse, extreme dietary habits, multiple food allergies, extreme levels of physical or athletic activity, or by changes in body weight >20 lbs. during the last 6 months
* Current use of antibiotics or during the previous 4 weeks.
* Inability to follow any of the experimental diets (including being vegetarian) or to perform the sampling required for this study
* Use of herbal supplements that may alter the gut microflora
* Autoimmune diseases
* Recent colonoscopy (within the previous two months)
* Use of antidiarrheal medication
* Thyroid diseases
* Use of omega-3 supplements (unless it is discontinued one month prior to the beginning of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
tryptophan metabolism | 1 week per intervention arm
  The response of plasma metabolites related to tryptophan metabolism to diets differing in saturated fat and prebiotics content (animal-based diet versus plant-based diet) will vary in individuals carrying CC (n=20) and TT (n=20) genotypes at the common APOA2 -265T>C single nucleotide polymorphism (SNP)

SECONDARY OUTCOMES:
Satiety assessment using plasma levels of leptin | 1 week per intervention arm
  Plasma leptin (ng/ml) will be measured in plasma during each one of the intervention phases. The response of leptin (ng/ml) to a saturated fat rich diet will be less on subjects with the CC genotype at the APOA2 locus as compared to TT subjects
adipose tissue metabolism | 1 week per intervention arm
  Plasma adiponectin (micrograms/ml) will be measured in plasma during each one of the intervention phases. The response of adiponectin to a saturated fat rich diet will be less on subjects with the CC genotype at the APOA2 locus as compared to TT subjects
Plasma Lipoproteins | 1 week per intervention arm
  Plasma lipoprotein concentrations in mg/dl (VLDL, LDL, HDL) and subclasses assessed by proton nuclear magnetic resonance (NMR) spectroscopy
Gut microbiota diversity and composition | 1 week per intervention arm
  A low saturated fat (SFA)/high prebiotic (plant-based) diet and a high SFA/low prebiotic (animal-based) diets have a differential effect on gut microbiota patterns according to the presence of the CC or TT genotypes at the APOA2-265T>C variant
Plasma levels of Interleukin 6 to assess inflammatory status | 1 week per intervention arm
  Plasma Levels of interleukin-6 (IL6) (pg/ml) will be measured during each of the dietary phases. IL6 will be higher in CC subjects at the APOA2 locus when consuming a high fat diet than when consuming a low fat diet. A low fat diet will not elicit increased IL6 levels in TT APOA2 subjects.
Plasma levels of tumor necrosis factor alpha to assess regulation of immune cells | 1 week per intervention arm
  Plasma Levels of tumor necrosis factor alpha (TNFA)(pg/ml) measured during each diet phase, will be significantly different depending on diet and APOA2 genotype. TNFA will be higher in CC subjects at the APOA2 locus when consuming a high fat diet than when consuming a low fat diet. A low fat diet will not elicit increased TNFA levels in TT APOA2 subjects.
Plasma levels of C-reactive to assess regulation of inflammation | 1 week per intervention arm
  Plasma Levels of C-reactive protein (CRP) (mg/L) measured during each diet phase will be significantly different depending on diet and APOA2 genotype. CRP will be higher in CC subjects at the APOA2 locus when consuming a high fat diet than when consuming a low fat diet. A low fat diet will not elicit increased CRP levels in TT APOA2 subjects.
Plasma levels of Lipopolysaccharides to assess gut inflammation | 1 week per intervention arm
  Plasma Levels of lipopolysaccharides (LPS) (ng/ml) will be significantly different depending on diet and APOA2 genotype. LPS will be higher in CC subjects at the APOA2 locus when consuming a high fat diet than when consuming a low fat diet. A low fat diet will not elicit increased LPS levels in TT APOA2 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Ordovas, PHD, Principal Investigator — JM-USDA HNRCA at Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corella D, Arnett DK, Tsai MY, Kabagambe EK, Peacock JM, Hixson JE, Straka RJ, Province M, Lai CQ, Parnell LD, Borecki I, Ordovas JM. The -256T>C polymorphism in the apolipoprotein A-II gene promoter is associated with body mass index and food intake in the genetics of lipid lowering drugs and diet network study. Clin Chem. 2007 Jun;53(6):1144-52. doi: 10.1373/clinchem.2006.084863. Epub 2007 Apr 19. PMID 17446329
- [Background] Corella D, Peloso G, Arnett DK, Demissie S, Cupples LA, Tucker K, Lai CQ, Parnell LD, Coltell O, Lee YC, Ordovas JM. APOA2, dietary fat, and body mass index: replication of a gene-diet interaction in 3 independent populations. Arch Intern Med. 2009 Nov 9;169(20):1897-906. doi: 10.1001/archinternmed.2009.343. PMID 19901143
- [Background] Smith CE, Tucker KL, Arnett DK, Noel SE, Corella D, Borecki IB, Feitosa MF, Aslibekyan S, Parnell LD, Lai CQ, Lee YC, Ordovas JM. Apolipoprotein A2 polymorphism interacts with intakes of dairy foods to influence body weight in 2 U.S. populations. J Nutr. 2013 Dec;143(12):1865-71. doi: 10.3945/jn.113.179051. Epub 2013 Oct 9. PMID 24108135